CLINICAL TRIAL: NCT04940728
Title: The Effect of an Intervention Program Based on Creative Thinking Techniques on the Problem Solving and Communication Skills of Nursing Students
Brief Title: Creative Thinking Problem Solving and Communication Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, YASEMİN ÖZEL, LECTURER, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KU-TOSYAMYO-YÖ-01
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Nursing Caries; Communication; Problem;Learning; Creativity
Keywords: Creativity; Creative thinking; Innovativeness,; Creative ability,; Education nursing; Problem solving skills; Communication skills
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: This research was designed in the experimental design model with pretest-posttest randomized control group, one of the quantitative research methods, in order to evaluate the effect of the intervention program developed based on creative thinking techniques on the problem solving and communication skills of nursing students.
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, the sample groups (experimental and control) were determined by an instructor other than the researchers, and the researchers were blinded while the sample was being created. The researchers and participants did not know who was in the experiment and who was in the control group during the assignment process until the study started. This method is a control method in which the participants in the study are blinded. After the assignment process took place, it was ensured that the students included in the research and the statistician evaluating the data did not know the experimental and control groups. In this context, two-way blinding method was used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creative Thinking Group (Experimental): Nursing students who took the Self-Knowledge and Communication Techniques course for the first time in March and agreed to participate in the study were divided into experimental (30) and control (30) groups using a simple randomization method.
  Pre-tests (Descriptive Information Form, Communication Skills Scale, and Problem Solving Scale) were administered to the participants who volunteered to participate in the research using the Online Questionnaire System.
  Considering the effect on the research data, after completing the routine courses of "self-knowledge", "communication skills", "listening skills" and "problem solving skills"; Intermediate tests (Communication Skills Scale, and Problem Solving Scale) were applied to the experimental and control groups.
  An intervention program based on creative thinking techniques was applied to the experimental group and post-tests (Communication Skills Scale, and Problem Solving Scale) were applied.
  Interventions: Other: Creative thinking techniques intervention program
- Standart Group (No Intervention): Pre-tests (Descriptive Information Form, Communication Skills Scale, and Problem Solving Scale) were applied to the participants who volunteered to participate in the study by using the Online Questionnaire System.
  Considering the effect on the research data, after completing the routine courses of "self-knowledge", "communication skills", "listening skills" and "problem solving skills" of the 4 main topics in the course; Intermediate tests (Communication Skills Scale, and Problem Solving Scale) were applied to the experimental and control groups by using the Online Questionnaire System.
  After the interim tests were applied, no intervention was made to the control group until the end of the period. At the end of the semester, post-tests (Communication Skills Scale, and Problem Solving Scale) were applied.

INTERVENTIONS:
Other: Creative thinking techniques intervention program — The intervention program based on creative thinking techniques was designed to consist of four stages: preparation, theoretical briefing, skill development and evaluation. In the first stage of the program, acquaintance and information meeting, in the second stage, the theoretical part lasts for two weeks, in the third stage, various creative thinking techniques are applied for four weeks to gain creative thinking skills.
  Arms: Creative Thinking Group

SUMMARY:
Creative thinking is a very important factor, especially due to recent developments in technology and health. In order to adapt and contribute to these developments, creativity is also very important for the nursing profession, which is a health discipline consisting of science and art. Creative thinking skills need to be developed so that nurses can develop healthy interpersonal relationships, find solutions to the problems they encounter in their working and social life, approach the patient with a holistic perspective, use the knowledge they have acquired in education life at an optimal level in the delivery of health services, produce new information and gain a critical perspective.

In today's information age, it is very important for professional development to develop the teaching models used in nursing education based on the philosophy of lifelong learning, to be revised frequently, to control the curriculum and to evaluate the effectiveness of the teaching techniques used at frequent intervals. The above-mentioned literature suggests that nurses should use creativity in their problem-solving and communication skills. In this context, it creates the need to use alternative creative thinking teaching techniques to develop nursing students' problem solving and communication skills. For this reason, the research was conducted to develop an intervention program based on creative thinking techniques in nursing education and to evaluate the effect of this program based on creative thinking techniques on problem solving and communication skills in nursing students. If a meaningful relationship is found between these variables and creative thinking education as a result of the research, the education program prepared on the subject will constitute a guide for the nursing curriculum in gaining creative thinking, problem solving and communication skills in nursing students.

DETAILED DESCRIPTION:
Thinking is a mental activity, one of the most important aspects of the learning process. The most important feature of the thinking process is that it does not involve action and is an action done before acting. In this context, the individual can evaluate the strategies he will choose to reach his goals by using his mental processes and imagination.

Creative thinking, one of the types of thinking, takes place in the first stage of the thinking process. At this stage, the person presents a new and original thought. In this context, it includes the skills to think creatively, generate new ideas, seek and find alternatives, adapt to a new approach, explore available options, and encourage assumptions. Creative thinking can be defined as shaping solutions to a problem or possible explanations of a phenomenon.

Creative thinking and problem solving actions are considered metacognitive processes within the scope of cognitive science. Cognition; It is defined as the formation of meta or meaningful knowledge from knowledge and thus the realization of learning. Metacognition is the executive and guiding mechanism that controls the thinking process within the scope of information processing. While the individual knows how he thinks and learns while using metacognitive information, he can plan, monitor and evaluate this process with metacognitive control. Therefore, metacognition has an important place in creative thinking skills. The most important reason for this is that creativity is a new and valuable thought development process.

Creative thinking is accepted as one of the core competencies of the twenty-first century and can be developed through education. Focusing on innovation draws attention to the need to develop creative thinking skills both in education and in other sectors. In this direction, the importance of developing creative thinking in nursing education emerges.

Creativity in nursing education is an important factor in teaching creative thinking, awareness level, interpersonal relations and problem solving skills for skill acquisition. The role of the education system is very important in the development of educational programs that will help develop students' creativity. It is seen that there are theorists emphasizing the importance of creativity directly or indirectly in nursing science. In this context, creative thinking can be beneficial in raising the individual's awareness level, developing healthy interpersonal relationships, finding a solution to a problem in relationships, and using the knowledge acquired during undergraduate education at an optimal level in the delivery of health services.

Learning communication skills, which is an important factor especially in psychiatric nursing, takes place primarily during undergraduate education. In this process, it is aimed to develop students personally and professionally both in theoretical courses and in practical training (clinical/field). When the studies on creative thinking are examined, it is seen that there are studies showing that creativity can be developed through education. Since the intervention program developed based on creative thinking techniques is thought to have an effect on the problem solving and communication skills of nursing students, the study was planned for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Not having a neurological problem
* Being able to communicate in Turkish mother tongue,
* To have active education in the nursing program
* To have taken the self-knowledge and communication course for the first time
* Volunteering to participate in the research

Exclusion Criteria:

* Be under the age of 18,
* Not having internet access
* Not being able to communicate in Turkish in mother tongue or being a foreign national,
* Have any previous training in creativity,
* Not volunteering to participate in the research,
* No internet use during the application process

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Communication Skills Scale | Four Months
  Communication Skills Inventory is a 5-point Likert-type Scale consisting of 45 items prepared in order to determine the communication skills levels of individuals. The items are (1) always, (2) usually, (3) sometimes, (4) rarely, and (5) never.
  The lowest score that can be obtained from the inventory is 45, and the highest score is 225. Each of the sub-dimensions consists of 15 items, including mental (Z) (1, 3, 6, 12, 15, 17, 18, 20, 23, 24, 26, 28, 33, 37 and 45), emotional (D) (5, 9, 11, 27, 29, 31, 34, 35, 36, 38-40 and 42-44), and behavioral (T) (2, 4, 7, 8, 10, 13) , 14, 16, 19, 21, 22, 25, 30, 32 and 41) measures communication skills. The higher the participant's sub-dimension score, the better his or her skill in that sub-dimension is interpreted. The high overall score is interpreted as being high in direct proportion to the communication skill.

SECONDARY OUTCOMES:
Problem Solving Scale | Four Months
  The Problem Solving Scale was developed in 1982 to determine how an individual perceives himself/herself regarding problem-solving behaviors and stages. It consists of 35 items: (1) always, (2) often, (3) often, (4) occasionally. , (5) rarely, (2) I never act like this is a 6-point Likert-type inventory.
  In the problem solving inventory, each question is given a score between 1 and 6. Inventory items consist of positive and negative judgments about problem solving and are arranged randomly. In scoring, negative items are evaluated with the reverse scoring method. Items 9, 22, 29 are not scored, and questions 1, 2, 3, 4, 11, 13, 14, 15, 17, 21, 25, 26, 30 and 34 are evaluated with the reverse scoring method. In the scoring of the inventory, the lowest 32 and the highest 192 points can be obtained. The high total scores obtained from the scale mean that the individual perceives himself as inadequate in terms of problem solving skills.

CONTACTS AND LOCATIONS:
Overall Officials: Birgül ÖZKAN, Assoc. Prof., Study Director — Ankara Yıldırım Beyazıt University Faculty of Health Sciences
Locations (1):
- Ankara Yıldırım Beyazıt University Faculty of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No